CLINICAL TRIAL: NCT03993444
Title: Prevent Pain and Stress Related Sickleave.
Acronym: PS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOT
Record Dates: First submitted 2019-05-29; First posted 2019-06-20 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stress, Psychological; Pain
MeSH Terms: conditions — Stress, Psychological; Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants receive one of two active conditions. Outcome assessors are not part of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- communication and problem solving (Experimental): Three smal group sessions (separate for employees (length 2 hours each) and for supervisors (length 2,5 hours each)) focused on training communication and problem solving skills.
  Interventions: Behavioral: communication and problem solving
- psychoeducation (Active Comparator): Two, 1 hour, lectures, one on the topic of pain and one on the topic of stress (for employees and supervisors combined).
  Interventions: Behavioral: psychoeducation

INTERVENTIONS:
Behavioral: communication and problem solving — a program for supervisors and employees including skills training, validating communication, problem solving
  Arms: communication and problem solving
Behavioral: psychoeducation — lecture/course for supervisors and employees on risk factors and actions for people experiencing stress and/or pain
  Arms: psychoeducation

SUMMARY:
Problems with stress and pain are common reasons for long-term sick-leave, and need preventive interventions. This RCT builds on a successful previous project (see reference section), where a program involving the work place, the individual and occupational health care resulted in decreased sick-leave and healthcare visits and a higher quality of life as compared to TAU for individuals with musculoskeletal pain. This study will replicate and evaluate the mechanisms behind the involvement from the work place. According to the transdiagnostic model, problems with stress and pain are maintained by similar processes. Consequently, the study will be extended to include both problems, and it will be explored how a refined version of the program affects sick leave and work ability in the employees.

DETAILED DESCRIPTION:
Compared to the earlier study, this RCT will include:

1. A focused program targeting supervisors and employees
2. An active control group
3. An evaluation of the effects on both supervisor and employee
4. Knowledge on the mechanisms involved
5. Replication and extension of earlier findings

The project will produce knowledge about:

A procedure for identifying individuals at risk for sick-leave. The effects of a program targeting both workplace and individual to prevent problems with stress and pain.

The role of the supervisor in preventing sick-leave. Mechanisms linked to decreased levels of sick-leave.

ELIGIBILITY:
Inclusion Criteria:

* participating employee has self rated symptoms of stress and/or pain and supervisor also partakes in intervention
* employed at a workplace within Regionhälsans (occupational health care center) uptake area

Exclusion Criteria:

* pain and/or stress symptoms due to medical conditions
* severe psychiatric conditions
* full time sick leave

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
sick leave | 14 months
  days on sick leave based on register data
sick leave | 8 months
  days on sick leave based on self report

SECONDARY OUTCOMES:
stress symptoms | baseline, 2 months, 8 months
  change in perceived stress scale-10, assessed in employees and supervisors
work ability | 2 months, 8 months
  work ability index, assessed in employees and supervisors
exhaustion symptoms | baseline, 2 months, 8 months
  change in Karolinska Exhaustion Disorder Scale, assessed in employees and supervisors
pain problems | baseline, 2 months, 8 months
  change in Örebro Musculoskeletal Pain Screening Questionaire, assessed in employees
work related factors | 2 months, 8 months
  QPS nordic, assessed in employees and supervisors
work limitations | 2 months, 8 months
  Work Limitations Questionnaire, assessed in employees
symptom catastrophizing | baseline, 2 months, 8 months
  change in Symptom Catastrophizing Scale, assessed in employees
problem framing | baseline, 2 months, 8 months
  change in Pain/stress Solutions questionnaire (PaSol), assessed in employees
communication | baseline, 2 months, 8 months
  change in Validation Invalidation Response Scale, assessed in employees
life satisfaction | 2 months, 8 months
  Brunnsviken Brief Quality of Life scale, assessed in employees and supervisors
health | 2 months, 8 months
  Visual Analogue Scale (0-100, higher values better health), assessed in employees and supervisors
communication behavior | baseline, 2 months
  change in Validating and Invalidating Behavior Coding Scale (VIBCS, two 0-7 scales, higher scores indicate higher levels of validating and invalidating communication)

OTHER OUTCOMES:
intervention credibility | baseline
  participant perception of intervention credibility, one item taken from the Credibility and expectancy questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: ida flink, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Center for Health and Medical Psychology (CHAMP) Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linton SJ, Boersma K, Traczyk M, Shaw W, Nicholas M. Early Workplace Communication and Problem Solving to Prevent Back Disability: Results of a Randomized Controlled Trial Among High-Risk Workers and Their Supervisors. J Occup Rehabil. 2016 Jun;26(2):150-9. doi: 10.1007/s10926-015-9596-z. PMID 26202039